CLINICAL TRIAL: NCT04125875
Title: Gastric Slow Wave and Autonomic Nervous Function in Cirrhotic Patients With
Brief Title: Gastric Slow Wave and Autonomic Nervous Function in Cirrhotic Patients With Esophageal Varices After Ligation-A Clinical Research
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-SR-086
Record Dates: First submitted 2019-08-05; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-08

CONDITIONS: Esophageal Varices in Cirrhosis of the Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cirrhosis of esophageal varices
  Interventions: Diagnostic Test: Electrogastrogram(EGG); Diagnostic Test: Heart Rate Variability(HRV)
- Patients with gastric polyps
  Interventions: Diagnostic Test: Electrogastrogram(EGG); Diagnostic Test: Heart Rate Variability(HRV)

INTERVENTIONS:
Diagnostic Test: Electrogastrogram(EGG) — Heart Rate Variability
Diagnostic Test: Heart Rate Variability(HRV) — Heart Rate Variability

SUMMARY:
This study is intended to include 20 patients with esophageal varices caused by liver cirrhosis who were admitted to the first affiliated hospital of nanjing medical university from May 2019, and randomly select 8 patients with gastric polyps as the control group.General clinical data, imaging data, endoscopic data and laboratory indicators were collected.Electrogastrogram (EGG) and Heart Rate Variability (HRV) were performed before and 24 hours after operation in patients with cirrhotic esophageal varices, and the dyspepsia scale was filled out.Electrogastrogram (EGG) and cardiac variability (HRV) were performed in patients with gastric polyps 24 hours before and after surgery, and the dyspepsia scale was filled.EGG uses the surface electrode to record gastric myoelectric activity, and evaluates the patient's gastric rhythm by normal slow wave ratio, overspeed ratio, overslow ratio, and rhythm disorder ratio.The HRV evaluates the balance state of the patient's autonomic nervous system with High Frequency (HF)/Low Frequency (LF).SPSS software was used for paired sample analysis of experimental results.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with cirrhosis of esophageal varices who underwent endoscopic ligation
* Signed informed consent

Exclusion Criteria:

* Hemorrhage in the digestive tract, unstable vital signs
* Hepatic encephalopathy
* Unwilling to cooperate with the examiner
* Skin allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with cirrhotic esophageal varices who were admitted to the First Affiliated Hospital of Nanjing Medical University since May 2019. Eight patients with gastric polyps were randomly selected as controls.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Gastric Slow Wave of patients before the surgery, Change from Baseline Gastric Slow Wave 1 day after the surgery ,Change from Baseline Gastric Slow Wave 5 days after the surgery | before the surgery, 1 day after the surgery, and 5 days after surgery
  EGG evaluate patient's gastric electrical rhythm by normal slow wave ratio, overspeed ratio, overslow ratio, and rhythm disorder ratio Evaluating patient's gastric electrical rhythm by normal slow wave ratio, overspeed ratio, overslow ratio, and rhythm disorder ratio Evaluating patient's gastric electrical rhythm by normal slow wave ratio, overspeed ratio, overslow ratio, and rhythm disorder ratio Evaluating patient's gastric electrical rhythm by normal slow wave ratio, overspeed ratio, overslow ratio, and rhythm disorder ratio

SECONDARY OUTCOMES:
LF/HF of patients before the surgery, Change from Baseline LF/HF 1 day after the surgery ,Change from Baseline LF/HF 5 days after the surgery | before the surgery, 1 day afterthe surgery, and 5 days after surgery
  HRV assesses the balance of the patient's autonomic nervous system with high frequency (HF) / low frequency (LF)

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Nanjing Medical Universit, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided